CLINICAL TRIAL: NCT07323316
Title: Holistic Assessment and Remote Digital MONitoring of mYasthenia Gravis Via MyoSense 360
Acronym: HARMONY 360
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADS-HARMONY360-2025
Record Dates: First submitted 2025-11-19; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MyoSense 360 (Experimental): Performance of digital tests (only at D0), digital questionnaires and standard test in clinic at D0, D180 and D360 Use of MyoSense 360 at-home in between visits during 12 months of follow-up and answer ePRO
  Interventions: Device: MyoSense 360

INTERVENTIONS:
Device: MyoSense 360 — The investigational version of MyoSense 360 consists of two mobile applications running on the patient's smartphone (CentrePoint Connect and InClinical), an ActiGraph LEAP activity monitor (Ametris product), as well as two cloud computing platforms

SUMMARY:
The purpose of the HARMONY 360 investigation is to explore the feasibility of using MyoSense 360 digital measures to develop models capable of detecting clinically meaningful changes in generalized Myasthenia Gravis (gMG) trajectory over 12 months under real-world conditions. Its main objective is not yet to demonstrate the final conformity of the device (exploratory study under article 82), but to collect preliminary data of safety and clinical performance that will help to refine the final product and inform the subsequent pivotal study.

The primary objective focuses on developing models to detect disease trajectory changes defined by the clinically significant +/- 2 points MG-ADL threshold. Secondary objectives include assessing usability, adherence, and the feasibility of models for worsening/exacerbation prediction. Finally, risks and anticipated Adverse Device Effects (ADEs) associated with the device use will be monitored continuously throughout the investigation. Consistent with its Proof of Concept stage, the study defines no claims of clinical performance, effectiveness or safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at screening
* Patients with gMG diagnosis confirmed by the investigator based at least on one of the following:
* Positive antibody testing for ACHR or MuSK antibodies; or,

  * LRP-4 antibodies or seronegative patients with additional positive single fiber examination; or,
  * Abnormal single-fiber EMG (SFEMG) jitter in at least one clinically weak muscle; or,
  * Objective evidence of improvement of clinical gMG symptoms following treatment with oral AChEI or positive pyridostigmine or neostigmine or edrophonium test
* MGFA Class IIa to IVb
* Having read the information sheet and signed the informed consent form
* Owning and able to use a personal smartphone which software version is above 16 for iOS and 8 for Android included
* Able to read languages in which the mobile application is available and able to understand pictograms (MyoSense 360 is available in local official languages)
* Able to use an activity monitor (per Actigraph LEAP activity monitor wearability criteria; see vendor guidance)
* For France only, affiliated with or benefiting from a social security system

Exclusion Criteria:

* Known medical or psychological condition(s) or risk factor(s) that, as judged by the investigator, might interfere with the subject's full participation in the study, pose any additional risk for the subject, or confound the assessment of the subject or outcome of the study.
* Person under guardianship or curatorship
* Current drugs or/and alcohol abuse that could influence performance on the tests, as judged by the investigator
* Participant has participated in another interventional clinical study within 30 days prior to screening or who are currently enrolled in another study that, in the - Investigator's opinion, could interfere with their full participation in this study or confound the assessment of the subject or study outcomes
* For France only, participant who has received more than €6,000 in compensation over the past 12 months for participating in human research, clinical trials, clinical investigations or performance studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To explore the feasibility of using digital measures collected by MyoSense 360 to develop models to detect changes in disease trajectory in adults with generalized Myasthenia Gravis over a 12-month period, under real-life, unsupervised conditions. | 12 months
  The primary endpoint will be the ability of the model to detect changes categorized as a 3-class variable:
  * improved: decreased Myasthenia Gravis Activities of Daily Living (MG-ADL) total score ≥2 points
  * unchanged: increased or decreased MG-ADL total score <2 points
  * worsening: increased MG-ADL total score by ≥2 points

SECONDARY OUTCOMES:
To explore the feasibility of using digital measures collected by MyoSense 360 to develop models to predict sustained worsening within a one-month forward-looking window | 1 month
  The first secondary endpoint will be the ability of the model to detect changes categorized as a 2-class variable:
  * worsening: increased MG-ADL total score by ≥2 points
  * other: either decreased MG-ADL total score ≥2 points or increased or decreased in MG-ADL total score <2 points
To describe the association between MyoSense 360 active functional tests combined measures in a model, obtained at home, without supervision and the standard reference QMG sub-items scores performed under clinical supervision at baseline. | 4 weeks
  Feasibility of using MyoSense 360 developed models to predict sustained worsening, i.e., an increase by at least 2-points in MG-ADL total score that is sustained within the next 4 weeks (no change observed in the opposite direction) will be described through performance metrics:
  - Positive predictive value
To describe the association between MyoSense 360 active functional tests combined measures in a model, obtained at home, without supervision and the standard reference QMG sub-items scores performed under clinical supervision at baseline. | 4 weeks
  Feasibility of using MyoSense 360 developed models to predict sustained worsening, i.e., an increase by at least 2-points in MG-ADL total score that is sustained within the next 4 weeks (no change observed in the opposite direction) will be described through performance metrics:
  - time-to-event accuracy
To describe the association between MyoSense 360 active functional tests combined measures in a model, obtained at home, without supervision and the standard reference QMG sub-items scores performed under clinical supervision at baseline. | 4 weeks
  Feasibility of using MyoSense 360 developed models to predict sustained worsening, i.e., an increase by at least 2-points in MG-ADL total score that is sustained within the next 4 weeks (no change observed in the opposite direction) will be described through performance metrics:
  - Model robustness across patients.
To describe the association between MyoSense 360 active functional tests measures obtained at home without supervision and the standard reference Quantitative Myasthenia Gravis (QMG) sub-items performed under clinical supervision at baseline | Day 0 and Day 1
  A correlation coefficient will be used to assess the relationship between the MyoSense 360 active functional tests at Day 1 (D1, at home) and standard tests at Day 0 (D0, in clinic). The endpoint will be considered positive if one test meets the expected correlation, with a minimum correlation threshold of r = 0.50 for the following comparisons:
  * "My Eyelids" Test (MET) and ptosis in QMG
  * "My Voice" Test (MVT) and onset of dysarthria in QMG
  * "My Breathing" Test (MBT) and vital capacity in QMG
  * "My Arms" test (MAT) and upper limb weakness in QMG
  * "My Legs" Test (MLT) and lower limb weakness in QMG
To describe the association between digital measures from MyoSense 360 (ActiGraph LEAP data collection, active smartphone functional tests and electronic Patient-Reported Outcomes) and clinical and patient-reported outcome measures | 12 months
  Cross-sectional and longitudinal associations between MyoSense 360 digital measures and clinical and patient-reported outcomes measured through questionnaires will be described using mixed-models
To describe participant compliance to the use of the MyoSense 360, including ActiGraph LEAP data collection all along the study, number of active functional tests performed and ePROs completed | 12 months
  Compliance to MyoSense 360 will be described through:
  - The number of days with valid* data collection from the wearable device.
  *The minimum requirement is 8 hours of daytime wear per day, with at least 60% daily compliance throughout the one-year follow-up period. Additionally, patients should wear the ActiGraph LEAP during at least two nights per week to capture relevant sleep and resting heart rate measures.
To describe the usability of MyoSense 360, including ActiGraph LEAP data collection, active functional tests and ePROs, from the patient's perspective. | Days 1, 180 and 345
  Usability of MyoSense 360 will be described using the System Usability Scale (SUS):
  - A descriptive analysis of the responses collected in the SUS related to the use of MyoSense 360 at Days 1, 180 and 345
To describe participant compliance to the use of the MyoSense 360, including ActiGraph LEAP data collection all along the study, number of active functional tests performed and ePROs completed | 12 months
  Compliance to MyoSense 360 will be described through:
  - The proportion of scheduled active functional tests completed per patient over time in comparison to the total expected
To describe overall patient satisfaction and perceived benefits of using MyoSense 360 in daily life | Days 1, 180 and 345
  Descriptive analysis of the answers collected in the patient's satisfaction and perceived benefits questionnaires related to the use of MyoSense 360
To monitor the incidence, type, and severity of adverse events and device deficiencies related to the use of MyoSense 360. | 390 days
  All adverse events (AEs), serious adverse events (SAEs) and Device Deficiencies (DD), and new findings on previous SAEs and DDs, suspected to be related to MyoSense 360 or not, will be prospectively collected from the first device use until 30 days after the last study activity, in line with ISO 14155:2020 and EU MDR 2017/745.